CLINICAL TRIAL: NCT01392651
Title: Outcome of Treatment of Women With Urinary Stress Incontinence Treated by Tension-free-vaginal-tape-obturator (TVTO) Compared to Tension-free-vaginal-tape-Secur (TVTS)
Brief Title: Tension-free-vaginal-tape-obturator (TVTO) Versus Tension-free-vaginal-tape-Secur (TVTS) for Treatment of SUI
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, menahem neuman, Principal Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: 920090039
Record Dates: First submitted 2011-06-27; First posted 2011-07-12 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2011-07

CONDITIONS: Urinary Stress Incontinence
Keywords: Urinary stress incontinence; TVT
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with urinary stress incontinence

SUMMARY:
Women with urinary stress incontinence who underwent surgical treatment by either TVTO or TVTS will be enrolled. The investigators will collect data from charts and use a telephone questionnaire to check the outcome of these women. Physical examination findings will also be incorporated.

ELIGIBILITY:
Inclusion Criteria:

* Women with USI who underwent TVTS or TVTO procedure, more than 6 months ago

Exclusion Criteria:

* Women who have not undergone TVT procedure

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with stress urinary incontinence who underwent surgery, by TVT methos, either TVTO or TVTS.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevention of stress incontinence | 12 months
  We will collect data from the files, question the women for possible urinary stress incontinence after one month, 6 months and 12 months after surgery. Data of physical examination will also be incorporated.

SECONDARY OUTCOMES:
Evaluation of side effects: tape erosion, pain, bleeding | 12 months
  We will question the women for possible pain, bleeding or vaginal discharge. The data on physical examination will be taken from the file.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Obstetrics and Gynecology, Western Galilee Hospital, Nahariya
  - Clinics of Dr Neuman, Rishon LeZiyyon